CLINICAL TRIAL: NCT03651375
Title: Hypofractionated 5x5 Gy Radiotherapy With Sequential Doxorubicin and Ifosfamide-based Chemotherapy in Marginally Resectable Soft Tissue Sarcomas of Extremities or Trunk Wall
Brief Title: Hypofractionated Radiotherapy With Sequential Chemotherapy in Marginally Resectable Soft Tissue Sarcomas of Extremities or Trunk Wall
Acronym: UN-RESARC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URESARC1
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Sarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Myosarcoma; Histiocytic Sarcoma; Synovial Sarcoma; Lymphangiosarcoma; Malignant Peripheral Nerve Sheath Tumors; Myxofibrosarcoma; Myxoid Liposarcoma; Undifferentiated Sarcoma; Pleomorphic Liposarcoma; Undifferentiated Pleomorphic Sarcoma; Dedifferentiated Liposarcoma; Pleomorphic Rhabdomyosarcoma; Malignant Triton Tumor
Keywords: Dose Hypofractionation; Neoadjuvant Therapy; Chemoradiotherapy; Sarcoma; Dose Fractionation; Dose-Response Relationship; Antineoplastic Agents; Drug Therapy; Antineoplastic Combined Chemotherapy Protocols
MeSH Terms: conditions — Sarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Myosarcoma; Histiocytic Sarcoma; Sarcoma, Synovial; Lymphangiosarcoma; Neurofibrosarcoma; Dermatofibrosarcoma; Liposarcoma, Myxoid; Histiocytoma, Malignant Fibrous | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sequential chemoradiotherapy (Experimental): 1xAI (doxorubicin 75 mg/sqm and ifosfamide 10 g/sqm) + 5x5 Gy radiotherapy + 2xAI + surgery
  Interventions: Drug: Sequential chemotherapy - 3 courses of AI; Radiation: Hypofractionated radiotherapy

INTERVENTIONS:
Drug: Sequential chemotherapy - 3 courses of AI — Three courses of doxorubicin and ifosfamide (AI, doxorubicin 75 mg/sqm and ifosfamide 10 g/sqm with prophylactic mesna), one before radiotherapy and two within the gap between radiotherapy and surgery.
Radiation: Hypofractionated radiotherapy — Preoperative hypofractionated 5x5 Gy radiotherapy (5 consecutive days) prescribed on planned target volume (tumor volume + elective margins + setup/error margin) with a daily image guidance with cone beam-CT-based position verification.

SUMMARY:
After a screening, which consists of biopsy, physical examination, initial diffusion-weighted magnetic resonance imaging (DWI-MRI), body computed tomography (CT) scan, blood tests and case analysis on Multidisciplinary Team (MDT) meeting, a patient will receive the first course of chemotherapy - doxorubicin 75 mg/sqm and ifosfamide 10 g/sqm (AI regimen) with prophylactic mesna. Then a patient will be irradiated 5x5 Gy and after radiotherapy he or she will receive two courses of AI within 4-6 weeks, depending on the tolerance. Then the response analysis in DWI-MRI and toxicity assessment and will be performed. On the second MDT meeting, a final decision about resectability of the tumor will be made. In case of resectability, a patient will be referred to surgery.

DETAILED DESCRIPTION:
There is lack of standard treatment of marginally resectable sarcomas. Results of commonly used approaches are unsatisfactory. The addition of neoadjuvant/induction chemotherapy before the irradiation and in the prolonged gap between the end of hypofractionated 5x5 Gy radiotherapy and surgery may allow to obtain the R0 resection rate, high pathological response rate and/or a higher rate of limb-sparing/conservative surgery as well as to increase patients' survival.

Hypofractionation represents a variation of radiotherapy fractionation in which the total dose is divided into fewer fractions with an increased fraction dose. Such treatment may lead to additional biological effects when compared to conventionally fractionated radiotherapy (eg. vascular damage, increased immunogenicity, and antigenicity). The main advantages of hypofractionation are those related to the decreased overall treatment time what is more convenient for both patients and physicians, increased compliance and makes the treatment more cost-effective. Intriguing, such an approach may provide an additional benefit when treating non-radiosensitive tumors with a low alpha/beta ratio (eg. sarcomas).

The basis of the study was a trial conducted by Kosela et al. in our center, which showed that preoperative short 5x5 Gy radiotherapy with immediate surgery is an effective and well-tolerated treatment of resectable sarcomas of extremities or trunk wall.

The rationale of chemotherapy comes from the interim analysis of a multicenter, international EORTC study comparing neoadjuvant systemic approaches in high-risk sarcomas. It was proven that AI regimen, which consists of ifosfamide and anthracyclines allowed to obtain 20% benefit in relapse-free survival and overall survival as compared to pathologically-tailored chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Age ≥18 years old
* Histologic diagnosis of soft tissue sarcoma
* Primary or recurrent tumor localized on extremities or trunk
* Grade 2 or grade 3 tumor
* Marginally resectable tumor as assessed by a multidisciplinary team
* Adequate renal function (serum creatinine ≤ 1.5 ULN)
* Adequate liver function (total bilirubin, AST, ALT 3x < ULN)

Exclusion Criteria:

* Radiation-induced sarcoma
* Second active malignancy, not including localized basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast; patients with a history of other malignancies are eligible if they have been continuously disease-free for > 10 years prior to the time of registration.
* History of radiation to the affected volume
* Histologic diagnosis of rhabdomyosarcoma (except pleomorphic subtype), angiosarcoma, epithelioid sarcoma, clear cell sarcoma, extraskeletal chondrosarcoma, alveolar soft part sarcoma, osteogenic sarcoma, Ewing's sarcoma/PPNET, aggressive fibromatosis, dermatofibrosarcoma protuberans
* Contraindications to radiotherapy, chemotherapy or surgery
* Metastatic disease except primary resectable isolated lung metastases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-02-11 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
The ratio of en limb-sparing/conservative R0 resections. | 24 months

SECONDARY OUTCOMES:
Radiological response in diffusion-weighted MRI | 24 months
  Radiological assessment of tumor change, especially diffusion parameters in DWI-MRI 6 weeks after the end of irradiation, according to the EORTC criteria.
Pathological response in resected tumors according to EORTC Soft Tissue and Bone Sarcoma Group criteria | 24 months
Toxicity of planned schedule of therapy according to CTCAE v.4.0. | 24 months after treatment completion
  The study will be stopped prematurely if the rate of non-hematological toxicity grade 3 >30%
2-years overall survival | 24 months after treatment completion
2-years local control rate | 24 months after treatment completion

OTHER OUTCOMES:
Assessment of biomarkers in biopsy and post-operative material | 24 months
  HIF-1 (hypoxia-inducible factor 1) - marker of hypoxia, predicting tumor response on radiotherapy; CD105/CD31/VEGF-A - tumor microvessel density; CD14, CD163, CD68KP i CD68 PG-M1 - tumor associated macrophages.

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Sklodowska-Curie Institute - Oncology Center, Warsaw, Mazovian, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barker HE, Paget JT, Khan AA, Harrington KJ. The tumour microenvironment after radiotherapy: mechanisms of resistance and recurrence. Nat Rev Cancer. 2015 Jul;15(7):409-25. doi: 10.1038/nrc3958. PMID 26105538
- [Background] Dumars C, Ngyuen JM, Gaultier A, Lanel R, Corradini N, Gouin F, Heymann D, Heymann MF. Dysregulation of macrophage polarization is associated with the metastatic process in osteosarcoma. Oncotarget. 2016 Nov 29;7(48):78343-78354. doi: 10.18632/oncotarget.13055. PMID 27823976
- [Background] Ellingsen C, Andersen LM, Galappathi K, Rofstad EK. Hypoxia biomarkers in squamous cell carcinoma of the uterine cervix. BMC Cancer. 2015 Oct 26;15:805. doi: 10.1186/s12885-015-1828-2. PMID 26502718
- [Background] Fujiwara T, Fukushi J, Yamamoto S, Matsumoto Y, Setsu N, Oda Y, Yamada H, Okada S, Watari K, Ono M, Kuwano M, Kamura S, Iida K, Okada Y, Koga M, Iwamoto Y. Macrophage infiltration predicts a poor prognosis for human ewing sarcoma. Am J Pathol. 2011 Sep;179(3):1157-70. doi: 10.1016/j.ajpath.2011.05.034. Epub 2011 Jul 21. PMID 21771572
- [Background] Ganjoo KN, Witten D, Patel M, Espinosa I, La T, Tibshirani R, van de Rijn M, Jacobs C, West RB. The prognostic value of tumor-associated macrophages in leiomyosarcoma: a single institution study. Am J Clin Oncol. 2011 Feb;34(1):82-6. doi: 10.1097/coc.0b013e3181d26d5e. PMID 23781555
- [Background] Gronchi A, Ferrari S, Quagliuolo, Broto M, J, Lopez-Pousa A, Grignani G, et al. Full-dose neoadjuvant anthracycline + ifosfamide chemotherapy is associated with a relapse free survival (RFS) and overall survival (OS) benefit in localized high-risk adult soft tissue sarcomas (STS) of the extremities and trunk wall: Interim analysis of a prospective randomized trial. Annals of Oncology, Volume 27, Issue suppl_6, 1 October 2016 https://academic.oup.com/annonc/article/27/suppl_6/LBA6_PR/2800561
- [Background] Jiang S, Yang Y, Fang M, Li X, Yuan X, Yuan J. Co-evolution of tumor-associated macrophages and tumor neo-vessels during cervical cancer invasion. Oncol Lett. 2016 Oct;12(4):2625-2631. doi: 10.3892/ol.2016.5014. Epub 2016 Aug 16. PMID 27698836
- [Background] Kim YH, Yoo KC, Cui YH, Uddin N, Lim EJ, Kim MJ, Nam SY, Kim IG, Suh Y, Lee SJ. Radiation promotes malignant progression of glioma cells through HIF-1alpha stabilization. Cancer Lett. 2014 Nov 1;354(1):132-41. doi: 10.1016/j.canlet.2014.07.048. Epub 2014 Aug 7. PMID 25109450
- [Background] Kosela-Paterczyk H, Szacht M, Morysinski T, Lugowska I, Dziewirski W, Falkowski S, Zdzienicki M, Pienkowski A, Szamotulska K, Switaj T, Rutkowski P. Preoperative hypofractionated radiotherapy in the treatment of localized soft tissue sarcomas. Eur J Surg Oncol. 2014 Dec;40(12):1641-7. doi: 10.1016/j.ejso.2014.05.016. Epub 2014 Sep 20. PMID 25282099
- [Background] Lee HJ, Yoon C, Park DJ, Kim YJ, Schmidt B, Lee YJ, Tap WD, Eisinger-Mathason TS, Choy E, Kirsch DG, Simon MC, Yoon SS. Inhibition of vascular endothelial growth factor A and hypoxia-inducible factor 1alpha maximizes the effects of radiation in sarcoma mouse models through destruction of tumor vasculature. Int J Radiat Oncol Biol Phys. 2015 Mar 1;91(3):621-30. doi: 10.1016/j.ijrobp.2014.10.047. Epub 2014 Dec 24. PMID 25544668
- [Background] Messiou C, Bonvalot S, Gronchi A, Vanel D, Meyer M, Robinson P, Morosi C, Bloem JL, Terrier PH, Lazar A, Le Pechoux C, Wardelman E, Winfield JM, Boulet B, Bovee J, Haas RL. Evaluation of response after pre-operative radiotherapy in soft tissue sarcomas; the European Organisation for Research and Treatment of Cancer-Soft Tissue and Bone Sarcoma Group (EORTC-STBSG) and Imaging Group recommendations for radiological examination and reporting with an emphasis on magnetic resonance imaging. Eur J Cancer. 2016 Mar;56:37-44. doi: 10.1016/j.ejca.2015.12.008. Epub 2016 Jan 20. PMID 26802529
- [Background] Wardelmann E, Haas RL, Bovee JV, Terrier P, Lazar A, Messiou C, LePechoux C, Hartmann W, Collin F, Fisher C, Mechtersheimer G, DeiTos AP, Stacchiotti S, Jones RL, Gronchi A, Bonvalot S. Evaluation of response after neoadjuvant treatment in soft tissue sarcomas; the European Organization for Research and Treatment of Cancer-Soft Tissue and Bone Sarcoma Group (EORTC-STBSG) recommendations for pathological examination and reporting. Eur J Cancer. 2016 Jan;53:84-95. doi: 10.1016/j.ejca.2015.09.021. Epub 2015 Dec 14. PMID 26700077
- [Background] Yehia L, Boulos F, Jabbour M, Mahfoud Z, Fakhruddin N, El-Sabban M. Expression of HIF-1alpha and Markers of Angiogenesis Are Not Significantly Different in Triple Negative Breast Cancer Compared to Other Breast Cancer Molecular Subtypes: Implications for Future Therapy. PLoS One. 2015 Jun 5;10(6):e0129356. doi: 10.1371/journal.pone.0129356. eCollection 2015. PMID 26046764
- [Background] Zhang M, Qiu Q, Li Z, Sachdeva M, Min H, Cardona DM, DeLaney TF, Han T, Ma Y, Luo L, Ilkayeva OR, Lui K, Nichols AG, Newgard CB, Kastan MB, Rathmell JC, Dewhirst MW, Kirsch DG. HIF-1 Alpha Regulates the Response of Primary Sarcomas to Radiation Therapy through a Cell Autonomous Mechanism. Radiat Res. 2015 Jun;183(6):594-609. doi: 10.1667/RR14016.1. Epub 2015 May 14. PMID 25973951